CLINICAL TRIAL: NCT07195708
Title: Clinical Study to Evaluate the Safety and Efficacy of the Orbera365 Intragastric Balloon System in Obese Patients
Brief Title: Orbera365 Intragastric Balloon System (Abbreviated as'Orbera365')
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E7236
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Experimental): Orbera365+Lifestyle management
  Interventions: Device: Treatment group
- Control group (No Intervention): Lifestyle management

INTERVENTIONS:
Device: Treatment group — The treatment group was the group with the placement of Orbera 365 plus lifestyle management
  Arms: Treatment group

SUMMARY:
To demonstrate the safety and efficacy of Orbera365 in obese populations to support the registration of Orbera365.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, randomized controlled, non-blinded trial.

The treatment group was the group with the placement of Orbera 365 plus lifestyle management, while the control group was the lifestyle management group. The central randomization system was adopted to randomly assign the research subjects into the experimental group and the control group. The subjects were enrolled at a 1:1 ratio, with 72 cases in each group, making a total of 144 cases.

The subjects in the treatment group will be followed up until 6 months after the balloon removal or 12 months after the endoscopy procedure, whichever comes later. The control group is planned to receive a 12-month lifestyle intervention, and the maximum follow-up period is up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is diagnosed with obesity, and the body mass index (BMI) is ≥28 kg/m² and ≤50 kg/m².
2. The subject is aged ≥18 years.
3. Failed previous conservative weight loss alternatives (e.g., supervised diet, exercise, and behavior modification programs).
4. Willing to avoid the use of medical devices, medications, or other substances for weight loss purposes during the study period.
5. Willing to avoid the use of nonsteroidal anti-inflammatory drugs (NSAIDs) during the study period, including aspirin, diclofenac, ibuprofen, naproxen, or other known gastric-irritating drugs.
6. Able to take proton pump inhibitors (PPIs), antiemetics, and other medications as prescribed by the researcher.
7. Capable of walking completely independently, with no severe chronic orthopedic diseases.
8. Willing to undergo gastroscopy.
9. Voluntarily participate in the trial, sign the informed consent form, and be willing to comply with study requirements, including follow-ups.

Exclusion Criteria:

1. Prior surgery involving the esophagus, stomach, and duodenum.
2. Prior bariatric surgery or intragastric medical devices for weight loss.
3. A large hiatal hernia of > 5 cm or a hernia ≤ 5 cm associated with severe or intractable gastroesophageal reflux symptoms.
4. Patients who have a history of gastrointestinal obstruction, adhesive peritonitis.
5. Any active inflammatory or neoplastic disease of the gastrointestinal tract. among these, inflammatory diseases include esophagitis, gastric ulcer, duodenal ulcer, and specific types (e.g., Crohn's disease), while neoplastic diseases include cancer, and the doctor judges that such conditions may affect the use of Orbera365.
6. Potential upper gastrointestinal bleeding disorders, such as esophageal or gastric varices, congenital or acquired intestinal capillary ectasia, or other congenital gastrointestinal abnormalities, such as atresia or stenosis that precludes the usage for Orbera365.
7. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope that precludes the usage for Orbera365.
8. Achalasia, symptoms suggestive of delayed gastric emptying, or presence of any other severe motility disorder that that may pose a safety risk during placement or removal of the device.
9. Positive result in the Helicobacter pylori breath test (Patients who turn negative after regular treatment can participate in this clinical trial).
10. History or symptoms of uncontrolled or unstable thyroid disease.
11. Abnormal coagulation with an INR > 1.5 that cannot be corrected (as judged by a physician) or requiring continuous full anticoagulant therapy, and/or the presence of any underlying disease associated with a high risk of bleeding.
12. Hepatic insufficiency or liver cirrhosis, including: acute liver failure, advanced liver cirrhosis with encephalopathy, muscle atrophy, and generalized edema. severe esophageal varices with red signs and gastric varices. severe portal hypertensive gastropathy with or without gastric antral vascular ectasia.
13. Anemia: For females, hemoglobin (Hgb) < 110 g/L. for males, hemoglobin (Hgb) < 120 g/L.
14. Patients with known or suspected allergic reactions to the materials contained in Orbera365.
15. Any other physical conditions that do not allow for elective endoscopy, such as poor overall health or a history and/or symptoms of severe kidney, liver, heart, and/or lung diseases. severe or uncontrolled mental illnesses or abnormalities that may affect the patient's ability to understand or comply with follow-up visits and the removal of the device 12 months later.
16. Patients who are unable or unwilling to take the prescribed proton pump inhibitor medications during the device placement period.
17. Patients who are unwilling to avoid any reconstructive and/or plastic surgeries that may affect weight during the study period, such as mammoplasty and liposuction.
18. Patients who are unwilling to participate in the established medical supervision diet and behavior modification program and undergo regular medical follow-ups.
19. Patients who are receiving treatment with anticoagulants, antiplatelet drugs, immunosuppressants, non-steroidal anti-inflammatory drugs (NSAIDs), or other drugs known to irritate the gastroduodenal mucosa or reduce gastrointestinal motility and/or are unwilling to discontinue such concomitant medications. prescription or over-the-counter weight loss drugs, drugs known to cause significant weight gain or loss (such as anesthetics, opioids, or benzodiazepines), insulin, antiepileptic drugs, antiarrhythmic drugs (such as amiodarone). other drugs that may cause weight changes, including drugs that can significantly increase weight (such as glucocorticoids, insulin secretagogues, thiazolidinediones, atypical antipsychotics, sodium valproate, lamotrigine, antidepressants, etc.), and drugs that can significantly reduce weight (such as glucagon-like peptide-1 receptor agonists, α-glucosidase inhibitors, topiramate, fluoxetine, bupropion, zonisamide, etc.).
20. Alcohol abuse and/or drug abuse.
21. Evidence of untreated mental or eating disorders, such as major depressive disorder, schizophrenia, substance abuse, binge eating disorder, or bulimia nervosa.
22. Poor overall health, presence of specific diseases, or situations that, in the judgment of the researcher during evaluation and/or device placement, may put the subject at significant risk, may confound the study results, may increase the risks associated with endoscopy and/or balloon placement, or may significantly interfere with the subject's participation in the study (for example, having acquired immunodeficiency syndrome or hepatitis C within the past 5 years).
23. Pregnant, breastfeeding, or having the intention to become pregnant during the study period (for females of childbearing potential).
24. Currently participating in a study of investigational drugs or devices, or having participated in such a study within 30 days before participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
%TBWL (Defined as the percentage of total body weight loss) | At 12 months after the intervention
  %TBWL is defined as the percentage of total body weight loss
The response rate at the 12th month after the intervention | At 12 months after the intervention
  Response is defined as having a percentage of total body weight loss (%TBWL) of ≥ 5%.